CLINICAL TRIAL: NCT00512317
Title: An Open-label Extension Study to Evaluate the Safety, Tolerability, and Efficacy of Ganaxolone as add-on Therapy in Adult Patients With Epilepsy Consisting of Uncontrolled Partial-onset Seizures.
Brief Title: Open-label Extension to Protocol 1042-0600
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1042-0601; V1.6
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Results first posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-12

CONDITIONS: Epilepsies, Partial
Keywords: partial onset epilepsy; adult epilepsy; partial seizures; anticonvulsant; catamenial epilepsy; adult partial onset epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Seizures | interventions — ganaxolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ganaxolone (Experimental): active experimental drug
  Interventions: Drug: ganaxolone

INTERVENTIONS:
Drug: ganaxolone — liquid suspension dosed tid

SUMMARY:
To allow open-label extension to patients who have completed Protocol 1042-0600.

DETAILED DESCRIPTION:
This is an open-label study evaluating efficacy and safety of ganaxolone treatment in adults with partial onset epilepsy with or without secondary generalizations.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have completed all scheduled clinical study visits in the previous protocol 1042-0600 and have been deemed eligible (no major adverse events thought to be drug related) by the Investigator.
2. Diagnosis of epilepsy with CPS with or without secondarily generalized seizures according to the International League Against Epilepsy [ILAE] Classification of Epileptic Seizures (1981). Diagnosis should have been established by clinical history and computerized tomography (CT) or magnetic resonance imaging (MRI) of the brain to rule out progressive structural lesions and electroencephalogram (EEG) or video EEG with results consistent with partial-onset epilepsy.
3. Male or female, 18 to 69 years of age (inclusive). [Note: Participants who are > 69 years of age but are of good health condition may be allowed to enter the study after discussion with and approval by the Medical Monitor.]
4. A 12-lead electrocardiogram (ECG) without clinically significant abnormalities.
5. Be properly informed of the nature and risks of the study and give informed consent in writing, prior to entering the study.
6. Able to participate for the full term of study.
7. Able to keep a seizure diary throughout the course of the study.
8. Sexually active women of childbearing potential must be using a medically acceptable method of birth control and have a negative qualitative serum beta-human chorionic growth hormone (beta HCG) pregnancy test result from a blood sample collected at the initial screening visit. A woman of childbearing potential is defined as a female who is biologically capable of becoming pregnant. A medically acceptable method of birth control includes intrauterine devices in place for at least 3 months, surgical sterilization, or adequate barrier methods (e.g., diaphragm and foam). An oral contraceptive alone is not considered adequate for the purpose of this study. Use of oral contraceptives in combination with another method (e.g., a spermicidal cream) is acceptable. In participants who are not sexually active, abstinence is an acceptable form of birth control and qualitative serum βHCG pregnancy tests must be tested per protocol.
9. Participants with a history of depression must be stable and may be taking one antidepressant medication

Exclusion Criteria:

1. Presence of non-motor simple partial seizures only.
2. History of pseudoseizures in the last 5 years.
3. History of a primary generalized seizure in the last 5 years.
4. Past use of vigabatrin without stable visual fields tested twice over the 12 months after the last dose of vigabatrin (Concomitant use of vigabatrin is not allowed).
5. Seizures secondary to illicit drug or alcohol use, infection, neoplasm, demyelinating disease, degenerative neurological disease, or CNS disease deemed progressive, metabolic illness, or progressive degenerative disease.
6. Status epilepticus within the last year prior to randomization in 1042-0600 study.
7. Clinically unstable psychiatric disorder within the last 2 years.
8. Suicide attempt within the last 5 years or current significant suicidal ideation.
9. History of psychosis within the last 5 years.
10. Current use of neuroleptics for psychosis.
11. A significant medical or surgical condition at screening which might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, or hepatic systems or other conditions that would place the participant at increased risk.
12. Known sensitivity or allergy to progesterone or related steroid compounds.
13. History of drug use or alcohol abuse within the past 5 years.
14. Sexually active women of childbearing potential (WCBP) who are unwilling to use a double-barrier method and establish that they are currently not pregnant by submitting to a serum pregnancy test.
15. A history of chronic noncompliance with drug regimens.
16. Females who are currently breastfeeding.
17. Exposure to any other investigational drug within 30 days prior to randomization in 1042-0600 study.
18. Aspartate transaminase (AST) or alanine transaminase (ALT) levels > 3 times the upper limit of normal (ULN) at screening.
19. Participant has history of repetitive seizures within the 12-month period preceding study entry where the individual seizures cannot be counted.
20. Inability to withhold grapefruit and grapefruit juice from diet during the entire clinical trial.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - University of Alabama, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Arkansas Epilepsy Program, Little Rock, Arkansas
  - University of Southern California Adult Comprehensive Epilepsy Center, Los Angeles, California
  - University of California-Davis, Sacramento, California
  - Anchutz Outpatient Pavillion Neurosciences Clinic/ University of Colorado Hospital, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida McKnight Brain Institute, Gainesville, Florida
  - Intercoastal Neurology, Sarasota, Florida
  - Emory HealthCare, Atlanta, Georgia
  - Southern Illinois University Medical Center, Springfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Dept. of Neurology, Lexington, Kentucky
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - 2799 West Grand blvd. CFP 071, Detroit, Michigan
  - Minnesota Epilepsy Group, PA, Saint Paul, Minnesota
  - Comprehensive Epilepsy Care Center for Children and Adults, Chesterfield, Missouri
  - Neurosciences Institute at Albany Medical Center, Albany, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Riddle Health Care Center for Neuroscience, Media, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Neurological Clinic of Texas, P.A., Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the previous double-blind controlled trial (Protocol 1042-0600, NCT00465517) were enrolled in this study.
Groups:
- Ganaxolone: Participants were administered ganaxolone (GNX) dose which ranged from 600 milligrams per day (mg/day) to 1500 mg/day oral liquid suspension. The dose titration schedule started with 300 mg three times daily (tid) (900 mg/day) and increased every 2 days by 100 mg tid (300 mg/day) to 500 mg tid (1500 mg/day). Participants who were able to tolerate the starting dose of 900 mg/day, were moved to increase dose of 1200 mg/day for 2 days, and then to 1500 mg/day until the optimal dose for efficacy and tolerability was achieved.
Period: Overall Study
Arm/Group | Ganaxolone
Started | 123
Completed | 6
Not Completed | 117
Not completed — Insufficient clinical response | 36
Not completed — Withdrawal by Subject | 23
Not completed — Sponsor closure of study | 21
Not completed — <50% reduction in seizure frequency on or after Visit 7 | 18
Not completed — Adverse Event | 13
Not completed — Discretion of the investigator or sponsor | 2
Not completed — Lost to Follow-up | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Groups:
- Ganaxolone: Participants were administered GNX dose which ranged from 600 mg/day to 1500 mg/day oral liquid suspension. The dose titration schedule started with 300 mg three times daily (tid) (900 mg/day) and increased every 2 days by 100 mg tid (300 mg/day) to 500 mg tid (1500 mg/day). Participants who were able to tolerate the starting dose of 900 mg/day, were moved to increase dose of 1200 mg/day for 2 days, and then to 1500 mg/day until the optimal dose for efficacy and tolerability was achieved.
Arm/Group | Ganaxolone
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.4 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 114
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 107
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Weekly Seizure Frequency During Weeks 1 Through 117
Description: Percent Change in weekly seizure frequency by treatment group compared to Baseline at the beginning of the double-blind study 1042-0600 is presented. Weekly seizure frequency included partial-onset seizures (POS) with or without secondary generalization, but not non-motor simple partial seizure (SPS) during Weeks 1 through Week 117. Baseline was defined as the Day 0 assessment before study drug infusion of the double-blind study 1042-0600.
Time Frame: Baseline (Day 0) and Week 1 through Week 117
Population: Intent-To-Treat (ITT) Population included all participants who received at least 1 dose of open-label study medication. Only participants who received at least 1 dose of ganaxolone in the open-label (OL) study (1042-0601), had seizure diary data for Baseline (from double-blind study 1042-0600), and who had data from at least 7 seizure diaries in the open-label study (1042-0601) were included. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- GNX/GNX: Ganaxolone in 1042-600 followed by Ganaxolone in Extension Study
- PBO/GNX: Placebo (PBO) In 1042-600 followed by Ganaxolone in Extension Study
Arm/Group | GNX/GNX | PBO/GNX
Number analyzed (Participants) | 79 | 41
Percent Change
  Weeks 1-10 | -14.8 (54.86) | -12.3 (64.08)
  Weeks 1-13 | -14.0 (52.91) | -13.7 (65.60)
  Weeks >13-26: number analyzed (Participants) | 50 | 31
  Weeks >13-26 | -19.6 (42.38) | -19.8 (56.43)
  Weeks >26-39: number analyzed (Participants) | 31 | 21
  Weeks >26-39 | -37.7 (33.79) | -48.6 (37.54)
  Weeks >39-52: number analyzed (Participants) | 28 | 19
  Weeks >39-52 | -29.1 (51.26) | -42.9 (59.81)
  Weeks >52-65: number analyzed (Participants) | 22 | 15
  Weeks >52-65 | -29.9 (51.85) | -43.1 (59.45)
  Weeks >65-78: number analyzed (Participants) | 16 | 13
  Weeks >65-78 | -41.4 (38.21) | -67.7 (23.09)
  Weeks >78-91: number analyzed (Participants) | 8 | 7
  Weeks >78-91 | -38.8 (66.24) | -43.6 (37.60)
  Weeks >91-104: number analyzed (Participants) | 4 | 1
  Weeks >91-104 | -69.4 (43.96) | -100 (NA) — Standard deviation could not be calculated as a single participant was analyzed
  Weeks >104-117: number analyzed (Participants) | 1 | 0
  Weeks >104-117 | -93.3 (NA) — Standard deviation could not be calculated as a single participant was analyzed |

2. Secondary Outcome: Number of Responders During Weeks 1 Through 117
Description: Responders were defined as participants experiencing ≥50% of reduction in mean weekly seizure frequency from the Baseline. Baseline was defined as the Day 0 assessment before study drug infusion of the double-blind study 1042-0600.
Time Frame: Baseline (Day 0) and Week 1 through Week 117
Population: ITT Population. Only subjects who received at least 1 dose of ganaxolone in the open-label study (1042-0601), had seizure diary data for Baseline (from double-blind study 1042-0600), and who had data from at least 7 seizure diaries in the open-label study (1042-0601) were included. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- PBO/GNX: Placebo In 1042-600 followed by Ganaxolone in Extension Study
Arm/Group | GNX/GNX | PBO/GNX
Number analyzed (Participants) | 79 | 41
Participants
  Weeks 1-10 | 22 | 11
  Weeks 1-13 | 19 | 12
  Weeks >13-26: number analyzed (Participants) | 50 | 31
  Weeks >13-26 | 12 | 8
  Weeks >26-39: number analyzed (Participants) | 31 | 21
  Weeks >26-39 | 11 | 12
  Weeks >39-52: number analyzed (Participants) | 28 | 19
  Weeks >39-52 | 10 | 10
  Weeks >52-65: number analyzed (Participants) | 22 | 15
  Weeks >52-65 | 8 | 8
  Weeks >65-78: number analyzed (Participants) | 16 | 13
  Weeks >65-78 | 6 | 11
  Weeks >78-91: number analyzed (Participants) | 8 | 7
  Weeks >78-91 | 4 | 4
  Weeks >91-104: number analyzed (Participants) | 4 | 1
  Weeks >91-104 | 3 | 1
  Weeks >104-117: number analyzed (Participants) | 1 | 0
  Weeks >104-117 | 1 |

3. Secondary Outcome: Number of Seizure-free Days During Weeks 1 Through 117
Description: Average number of seizure-free days per week for a given period was calculated as follows: (Total number of days with no seizures of any type during that period / number of days with seizure diary in that period) multiplied by 7.
Time Frame: Week 1 through Week 117
Population: ITT Population. Only participants who received at least 1 dose of ganaxolone in the open-label study (1042-0601), had seizure diary data for Baseline (from double-blind study 1042-0600), and who had data from at least 7 seizure diaries in the open-label study (1042-0601) were included. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Seizure free days
Arm/Group | GNX/GNX | PBO/GNX
Number analyzed (Participants) | 79 | 41
Seizure free days
  Weeks 1-10 | 4.8 (1.99) | 5.0 (1.81)
  Weeks 1-13 | 4.8 (1.97) | 5.0 (1.85)
  Weeks >13-26: number analyzed (Participants) | 50 | 31
  Weeks >13-26 | 5.1 (1.54) | 5.3 (1.40)
  Weeks >26-39: number analyzed (Participants) | 31 | 21
  Weeks >26-39 | 5.2 (1.69) | 5.4 (1.75)
  Weeks >39-52: number analyzed (Participants) | 28 | 19
  Weeks >39-52 | 5.4 (1.66) | 5.4 (1.56)
  Weeks >52-65: number analyzed (Participants) | 22 | 15
  Weeks >52-65 | 5.1 (2.11) | 5.2 (2.10)
  Weeks >65-78: number analyzed (Participants) | 16 | 13
  Weeks >65-78 | 5.3 (1.93) | 5.7 (1.61)
  Weeks >78-91: number analyzed (Participants) | 8 | 7
  Weeks >78-91 | 5.4 (2.32) | 4.7 (1.88)
  Weeks >91-104: number analyzed (Participants) | 4 | 1
  Weeks >91-104 | 5.6 (2.56) | 6.8 (NA) — Standard deviation could not be calculated as a single participant was analyzed
  Weeks >104-117: number analyzed (Participants) | 1 | 0
  Weeks >104-117 | 6.9 (NA) — Standard deviation could not be calculated as a single participant was analyzed |

4. Secondary Outcome: Number of Seizure-free Participants
Description: Number of Seizure-free participants is presented.
Time Frame: Day 1 through Day 224 (Week 32)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GNX/GNX | PBO/GNX
Number analyzed (Participants) | 79 | 41
Participants
  >=1 day | 75 | 41
  >= 28 days (4 weeks): number analyzed (Participants) | 71 | 38
  >= 28 days (4 weeks) | 20 | 38
  >= 56 days (8 weeks): number analyzed (Participants) | 61 | 33
  >= 56 days (8 weeks) | 6 | 33
  >=70 days (10 weeks): number analyzed (Participants) | 55 | 31
  >=70 days (10 weeks) | 4 | 31
  >=91 days (13 weeks): number analyzed (Participants) | 50 | 29
  >=91 days (13 weeks) | 4 | 29
  >=119 days (17 weeks): number analyzed (Participants) | 45 | 27
  >=119 days (17 weeks) | 43 | 27
  >=133 days (19 weeks): number analyzed (Participants) | 45 | 27
  >=133 days (19 weeks) | 3 | 27
  >=154 days (22 weeks): number analyzed (Participants) | 38 | 25
  >=154 days (22 weeks) | 3 | 25
  >=182 days (26 weeks): number analyzed (Participants) | 30 | 20
  >=182 days (26 weeks) | 0 | 20
  >=224 days (32 weeks): number analyzed (Participants) | 27 | 18
  >=224 days (32 weeks) | 0 | 18

5. Secondary Outcome: Change From Baseline in Quality of Life in Epilepsy Inventory-31 (QOLIE-31) Questionnaire
Description: QOLIE-31 was a survey of health-related QOL for adults with epilepsy and evaluated how much distress the participant feels about problems and worries related to epilepsy. It included 38 items grouped into eight multi-item subscales - Energy/Fatigue, Emotional Well-Being, Daily Activities/Social Functioning, Cognitive Functioning, Medication Effect, Seizure Worry, Overall Quality of Life (QoL) and Distress. The subscale scores and the total score were calculated according to the scoring algorithm defined by the author with scores ranging from 0 to 100; higher scores indicated better function. Baseline was defined as the last non-missing observation prior to the first dose in double-blind study 1042-0600. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 0) and up to Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | GNX/GNX | PBO/GNX
Number analyzed (Participants) | 42 | 18
Scores on a Scale
  Energy/Fatigue | -5.7 (18.16) | 3.9 (17.20)
  Emotional Well-Being | -4.7 (13.83) | 3.3 (22.13)
  Social Function | -3.6 (24.67) | 8.4 (21.44)
  Cognitive | 2.1 (19.91) | 2.9 (18.04)
  Medication Effect | -3.9 (25.28) | 0.9 (26.85)
  Seizure Worry | 3.6 (25.40) | -3.1 (35.73)
  Overall QoL | -3.8 (17.26) | 0.0 (15.17)
  Distress | -5.5 (18.49) | 0.7 (21.92)

ADVERSE EVENTS:
Time Frame: Up to Week 117
Description: AEs and SAEs were collected in ITT Population. No separate analysis was performed to report results by doses.
Groups:
- Ganaxolone: Participants were administered ganaxolone (GNX) dose which ranged from 600 mg/day to 1500 mg/day oral liquid suspension. The dose titration schedule started with 300 mg tid (900 mg/day) and increased every 2 days by 100 mg tid (300 mg/day) to 500 mg tid (1500 mg/day). Participants who were able to tolerate the starting dose of 900 mg/day, were moved to increase dose of 1200 mg/day for 2 days, and then to 1500 mg/day until the optimal dose for efficacy and tolerability was achieved.
Arm/Group | Ganaxolone
All-Cause Mortality (participants affected / at risk) | 0/123
Serious Adverse Events (participants affected / at risk) | 15/123
Other Adverse Events (participants affected / at risk) | 103/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=123)
Gastroenteritis salmonella (Infections and infestations) | 1
Convulsion (Nervous system disorders) | 7
Escherichia sepsis (Infections and infestations) | 1
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1
Pneumonia (Infections and infestations) | 1
Status epilepticus (Nervous system disorders) | 1
Cholelithiasis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 1
Osteomyelitis (Infections and infestations) | 1
Paraplegia (Nervous system disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Tooth abscess (Infections and infestations) | 1
Transaminases increased (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=123)
Anaemia (Blood and lymphatic system disorders) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac flutter (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Diplopia (Eye disorders) | 3
Vision blurred (Eye disorders) | 3
Asthenopia (Eye disorders) | 2
Ulcerative keratitis (Eye disorders) | 2
Blepharospasm (Eye disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Macular degeneration (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Oscillopsia (Eye disorders) | 1
Saccadic eye movement (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Stomach discomfort (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Hypoaestheisa oral (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Tongue disorders (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 20
Asthenia (General disorders) | 6
Pyrexia (General disorders) | 5
Gait disturbance (General disorders) | 4
Pain (General disorders) | 4
Irritability (General disorders) | 3
Non-cardiac chest pain (General disorders) | 3
Oedema peripheral (General disorders) | 2
Pitting oedema (General disorders) | 2
Facial pain (General disorders) | 1
Feeling abnormal (General disorders) | 1
Feeling drunk (General disorders) | 1
Influenza like illness (General disorders) | 1
Malaise (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Nasopharyngitis (Infections and infestations) | 17
Upper respiratory tract infection (Infections and infestations) | 10
Sinusitis (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 7
Bronchitis (Infections and infestations) | 3
Ear infection (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Localised infection (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Vulvovaginal mycotic infection (Infections and infestations) | 2
Candiduria (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis salmonella (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Trichomoniasis (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Vulval abscess (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 17
Contusion (Injury, poisoning and procedural complications) | 15
Skin laceration (Injury, poisoning and procedural complications) | 7
Excoriation (Injury, poisoning and procedural complications) | 3
Rib fracture (Injury, poisoning and procedural complications) | 3
Thermal burn (Injury, poisoning and procedural complications) | 3
Head injury (Injury, poisoning and procedural complications) | 2
Joint injury (Injury, poisoning and procedural complications) | 2
Joint sprain (Injury, poisoning and procedural complications) | 2
Limb injury (Injury, poisoning and procedural complications) | 2
Mouth injury (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1
Back injury (Injury, poisoning and procedural complications) | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1
Eye injury (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Weight increased (Investigations) | 2
Blood glucose increased (Investigations) | 1
Body temperature increased (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 1
Grip strength decreased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Urine analysis abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
White blood cells urine positive (Investigations) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Bunion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 26
Convulsion (Nervous system disorders) | 20
Dizziness (Nervous system disorders) | 16
Somnolence (Nervous system disorders) | 10
Nystagmus (Nervous system disorders) | 7
Coordination abnormal (Nervous system disorders) | 6
Balance disorder (Nervous system disorders) | 4
Sensory loss (Nervous system disorders) | 4
Cognitive disorder (Nervous system disorders) | 3
Amnesia (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Sedation (Nervous system disorders) | 2
Aphasia (Nervous system disorders) | 1
Complex partial seizures (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Hyposmia (Nervous system disorders) | 1
Intention tremor (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Postical state (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Status epliepticus (Nervous system disorders) | 1
Tongue paralysis (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Visual field defect (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 6
Abnormal dreams (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Stress (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 2
Affective disorder (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Thinking abnormal (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Leukocyturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Pyuria (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urine flow decreased (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 3
Menstruation irregular (Reproductive system and breast disorders) | 3
Breast tenderness (Reproductive system and breast disorders) | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 2
Breast mass (Reproductive system and breast disorders) | 1
Breast swelling (Reproductive system and breast disorders) | 1
Genital pruritus female (Reproductive system and breast disorders) | 1
Haematospermia (Reproductive system and breast disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Nipple pain (Reproductive system and breast disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngeal erthema (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 7
Ecchymosis (Skin and subcutaneous tissue disorders) | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Medical device change (Surgical and medical procedures) | 2
Brain lobectomy (Surgical and medical procedures) | 1
Sinus operation (Surgical and medical procedures) | 1
Uterine dilation and curettage (Surgical and medical procedures) | 1
Vasodilation procedure (Surgical and medical procedures) | 1
Hot flush (Vascular disorders) | 2
Flushing (Vascular disorders) | 1
Vein disorder (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No